CLINICAL TRIAL: NCT07141368
Title: An Open Label, Randomized, Balanced, Four-Treatment, Four-Sequence, Four-Period, Four-way Crossover, Single Oral Dose Comparative Bioavailability Study of Curcumin in Healthy Human Subjects Under Fasting Conditions.
Brief Title: Single Oral Dose Comparative Bioavailability Study of Investigational Product in Healthy Human Subjects Under Fasting Conditions.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 061-25
Record Dates: First submitted 2025-07-08; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: An Open Label, Randomized, Balanced, Four-Treatment, Four-Sequence, Four-Period, Four-way cross-over, Single Oral dose comparative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Curcumin Dispersome formulation (Experimental): 75% BLG (600 mg (2 capsules of 300 mg each, containing 90 mg curcumin per capsule
  Interventions: Other: Curcumin Dispersome formulation
- Non-formulated Curcumin (Experimental): dose: 90 mg, 1 capsule
  Interventions: Other: Non-formulated Curcumin
- Benchmark Formulation 1 - Turmipure Gold™ (Active Comparator): recommended daily dose: 300 mg, 1 capsule
  Interventions: Other: Benchmark Formulation 1 - Turmipure Gold™
- Benchmark Formulation 2 - Qunol, Turmeric, Curcumin Complex, Extra Strength (Active Comparator): recommended daily dose: 1000 mg, 2 capsules of 500 mg each
  Interventions: Other: Benchmark Formulation 2 - Qunol, Turmeric, Curcumin Complex, Extra Strength

INTERVENTIONS:
Other: Curcumin Dispersome formulation — 75% BLG (600 mg (2 capsules of 300 mg each, containing 90 mg curcumin per capsule
  Arms: Curcumin Dispersome formulation
Other: Non-formulated Curcumin — dose: 90 mg, 1 capsule
  Arms: Non-formulated Curcumin
Other: Benchmark Formulation 1 - Turmipure Gold™ — recommended daily dose: 300 mg, 1 capsule
  Arms: Benchmark Formulation 1 - Turmipure Gold™
Other: Benchmark Formulation 2 - Qunol, Turmeric, Curcumin Complex, Extra Strength — recommended daily dose: 1000 mg, 2 capsules of 500 mg each
  Arms: Benchmark Formulation 2 - Qunol, Turmeric, Curcumin Complex, Extra Strength

SUMMARY:
The sponsor has developed new curcuminoid formulations with the expectation of enhanced bioavailability compared to existing benchmark products. This study aims to evaluate the comparative bioavailability and characterize the pharmacokinetic profile of the test formulations in comparison to the reference formulations in healthy adult subjects under fasting conditions.

DETAILED DESCRIPTION:
This study is an open-label, randomized, balanced, single oral dose, four-treatment, four-sequence, four-period, four-way cross-over comparative bioavailability trial designed to assess the bioavailability of different curcumin formulations in healthy adult volunteers under fasting conditions. A total of 24 subjects will be enrolled, each receiving four investigational products in a randomized sequence: non-formulated curcumin (90 mg, 1 capsule), Curcumin Dispersome formulation (600 mg; 2 x 300 mg capsules, each containing 90 mg curcumin), Turmipure Gold™ (300 mg, 1 capsule), and Qunol, Turmeric, Curcumin Complex, Extra Strength (1000 mg; 2 x 500 mg capsules). Each product will be administered as a single oral dose with 240 mL of water after at least 10 hours of fasting. Subjects will be housed in the clinical facility for at least 36 hours prior to dosing and remain for at least 24 hours post-dose during each period, with a minimum 7-day washout between periods. Safety will be monitored through clinical examination, vital signs, ECG, and laboratory assessments throughout the study. Blood samples for pharmacokinetic analysis will be collected at 13 time points in each period, and subjects will receive standardized turmeric-free meals and adhere to strict dietary and medication restrictions. The primary objective is to compare the bioavailability of the investigational products, with secondary objectives including the evaluation of safety and tolerability in the study population.

ELIGIBILITY:
Inclusion Criteria:

* 9.5.1 Able and willing to participate in the study by complying with the protocol procedures as evidenced by a dated and signed informed consent form 9.5.2 Age greater than equal to 18 less than equal to 45 years. 9.5.3 Willing to consume the study product and donate blood. 9.5.4 BMI from 18.5 to 29.9 kg/m². 9.5.5 Subject with normal health as determined by personal medical and medication history, clinical examination and laboratory examinations within the clinically acceptable limits.

9.5.6 Subjects having vital parameters (blood pressure, body temperature, pulse rate and respiratory rate) within acceptable limits.

9.5.7 Non-smokers or mild/moderate smokers with not more than 10 bidis/cigarettes/pipes per day, and willing to abstain from smoking or chewing any tobacco containing products at least 72.00 hours prior to check-in and throughout the sampling points.

9.5.8 Agreeing not to consume food, drink and condiment containing curcumin (e.g. curry), or other curcuminoids (DMC, BDMC) for the whole duration of the study (36 hours pre-dose to 24 hours post-dose in each period).

9.5.9 Good general and mental health in the opinion of the investigator: no clinically significant or relevant abnormalities upon review of medical history or following a physical examination prior to check-in.

9.5.10 If study volunteer is a female and is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator, such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence Or She is surgically sterile (had a bilateral tubal ligation, bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 06 months).

Exclusion Criteria:

* 9.6.1 Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract or may affect absorption of IP and blood forming organ.

9.6.2 Significant history or current evidence of malignancy or chronic - infectious, cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic (endocrine), hematological, gastrointestinal, immunological or psychiatric disease or organ dysfunction.

9.6.3 Any major illness or hospitalization within 90 days prior to first admission to the study.

9.6.4 Use of any depot injection or an implant of any drug within 3 months prior to check-in and throughout the study.

9.6.5 Use of any prescribed medication or OTC (including herbal drugs and vitamin supplements) within 14 days prior to check-in and throughout the study.

9.6.6 Use of botanical dietary supplements during the study or within three months prior to check-in.

9.6.7 Difficulty in swallowing capsules. 9.6.8 History or presence of alcohol abuse in the past one year [Alcohol abuse will be defined as greater than 14 drinks per week (1 drink equal to 360 mL beer, 150 mL wine, or 45 mL hard liquor)].

9.6.9 Consumption of alcoholic products within 24.00 hours prior to check-in in each study period and throughout sampling time points.

9.6.10 Positive alcohol breath or urine drug of abuse test during check-in on each study period.

9.6.11 Consumption of xanthine's or its derivative containing food or beverages (e.g. chocolates, tea, coffee or cola drinks) within 48.00 hours prior to check-in and throughout sampling time points.

9.6.12 Consumption of grapefruit or its juice within 72.00 hours prior to check-in in each period and throughout sampling time points.

9.6.13 History of allergy or hypersensitivity intolerance to turmeric or curcumin.

9.6.14 Individuals who, in the opinion of the investigator, are unlikely to be able to comply with the study.

9.6.15 Irritable bowel syndrome. 9.6.16 Current disease states that are contraindicated with dietary supplementation: chronic diarrhea, constipation or abdominal pain, chronic laxatives use.

9.6.17 Pathology which could affect the study results or expose the subject to an additional risk according to the investigator.

9.6.18 Recent gastroenteritis or food borne illness such as confirmed food poisoning (less than 1 month).

9.6.19 Blood donation within 90 Days prior to the initial visit or intending to donate within the next 90 Days.

9.6.20 Low venous capital not allowing blood kinetic sampling. 9.6.21 Known or suspected food allergy, intolerance, or hypersensitivity to any of the study product ingredients and/or of the standard meals (gluten intolerance, celiac disease, etc.) 9.6.22 Chronic drug treatment (for example anticoagulant, antihypertensive medication, thyroid treatment, asthma treatment, anxiolytic, antidepressant, lipid-lowering treatment, corticosteroids, phlebotonic, veino-tonic, drug with impact on blood circulation) excluding oral and local contraceptives.

9.6.23 Currently taking (or during the past 3 months) any botanical dietary supplement.

9.6.24 History of anorexia nervosa, bulimia, or significant eating disorders according to the investigator.

9.6.25 Participation in another clinical trial 90 days prior to check-in period I of this study.

9.6.26 Presenting a psychological or linguistic incapability to sign the informed consent.

9.6.27 Female volunteer who has used implanted or injected hormonal contraceptives anytime during the 06 months prior to check-in or used hormonal contraceptives within 14 days before check-in

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of investigational products when compared with benchmark products, for Comparative Bioavailability Assessment (Cmax, AUC) under Fasting Conditions. | Pre-dose at -1.00 and 0.00 hours (within 10 minutes prior to dosing), and at 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 4.00, 6.00, 8.00, 12.00, and 24.00 hours post-dose.
  To assess the comparative bioavailability of investigational products versus benchmark products by evaluating pharmacokinetic parameters including maximum observed plasma concentration (Cmax) and area under the plasma concentration-time curve (AUC), in healthy adult subjects under fasting conditions.

SECONDARY OUTCOMES:
Number of Participants With safety and tolerability of the product after Administration of Curcumin | From pre-dose (-1.00 and 0.00 hours) to 24 hours post-dose (0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 4.00, 6.00, 8.00, 12.00, and 24.00 hours).
  The safety and tolerability of Curcumin will be evaluated by monitoring and recording, including physical examination findings, clinical laboratory results, vital signs, and participant-reported symptoms, following administration under fasting conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sanjay Vaze, MBBS, Principal Investigator — Vedic Lifesciences Pvt.Lts
Locations (1):
- IndiGlobal Labs Pvt. Ltd, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No